CLINICAL TRIAL: NCT01547065
Title: Use of Transesophageal Echocardiography to Measure Intraoperative Renal Resistive Index and Predict Acute Renal Injury
Status: Terminated | Type: Observational
Why Stopped: Enrollment lower than anticipated
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: 0120110047
Record Dates: First submitted 2012-03-02; First posted 2012-03-07 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Subjects Undergoing Cardiac or Major Surgery Where TEE is Used as a Matter of Routine
Keywords: TEE and renal resistive index

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators hypothesize that transesophageal echocardiography is a valid method to obtain renal doppler hemodynamics2, 4. The goal of this study is to determine if there is a correlation between abnormal TEE resistive index measurements, intraoperative events and post-operative creatinine changes

DETAILED DESCRIPTION:
The significant morbidity and mortality associated with acute kidney injury in critical care patients and after cardiac surgery is well-known. Studies have demonstrated between 1 to 30% postoperative mortality and even higher rates of up to 70% when patients develop renal failure and require dialysis. Even small increases in creatinine between 0 to 0.5 mg/dl can result in a greater than two-fold rise in 30-day mortality.1 Despite efforts to improve outcome, there has been no proven effective pharmacological interventions to treat acute kidney failure. Most recommendations are aimed at prevention by identifying high-risk patients, avoiding nephrotoxic drugs and minimizing intraoperative hypotensive insults.2

There are few studies that have examined the maintenance of adequate renal perfusion by measuring renal blood flow using transesophageal echocardiography (TEE) during cardiopulmonary bypass.3, 4 Yang et al. examined the left renal artery of 60 patients using TEE during cardiac surgery and evaluated the feasibility of using TEE as a method to measure renal blood flow intraoperatively.4 Although they were only able to include 60% of the subjects due to technical difficulties, they did demonstrate less than 10% variability between measurements and therefore good reproducibility using TEE. However, renal blood flow may not be the best method to predict sufficient renal perfusion. Renal autoregulation is not preserved under general anesthesia even with the maintenance of adequate mean arterial blood pressure and cardiac output. Renal blood flow is further worsened by hemodilution and hypothermia. In addition, due to its pulsatile nature, the diameters of the renal arteries vary during the cardiac cycle and are a source of calculation error when determining renal blood flow as a function of renal blood velocity and arterial diameter.2

Renal resistive index (RI) is a measure of intrarenal hemodynamics that is calculated using the blood flow velocities of segmental or intrarenal vessels and correlates with renal blood flow and renovascular resistance. The renal artery is not used because the flow varies and is inconsistent between systole and diastole. RI becomes elevated in pathological conditions and is associated with increasing creatinine, renal injury and dysfunction.5-7 As blood flow and creatinine clearance decrease through the renal vasculature, the resistive index increases. Resistive index may be a better gauge of renal dysfunction rather than renal blood flow because it is easier to assess and less dependent on obtaining a Doppler beam view that is oriented perfectly parallel to the blood flow.2 Because RI is a ratio of the renal blood flow velocities [RI = (peak systolic velocity - peak end diastolic velocity)/peak systolic velocity], the margin of error created by non-parallel Doppler beams cancels out.

Traditionally, resistive index is obtained by transabdominal Doppler ultrasonography (USG) although there have been transesophageal studies that have used RI as a secondary endpoint when examining renal blood flow.2, 4 There is currently no technique that routinely uses TEE to intraoperatively monitor resistive index as a determination of adequate renal blood perfusion and an indication of renal compromise.8 In addition, while other studies have reported RI as a secondary outcome, no studies have validated the TEE calculation of resistive index compared to the established transabdominal doppler technique.

ELIGIBILITY:
Inclusion Criteria:

* TEE is part of a anesthetic plan as determined by the anesthesiologist

Exclusion Criteria:

* Subjects on hemodialysis/peritoneal dialysis
* Subjects with a contraindication to use of TEE; esophageal stricture, esophageal diverticulum, esophageal tumor, recent esophageal/gastric surgery or radiation to the chest
* Subjects who are pregnant
* Subjects with esophageal varices
* Subjects with bleeding disorders

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: potential subjects are those undergoing cardiac or major abdominal or vascular surgery where TEE is standard of care
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2011-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
renal resistive index | intraoperatively

SECONDARY OUTCOMES:
post operative creatinine changes | 5 days post operatively
  subjects Blood Urea Nitrogen and creatinine levels will be recorded daily

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Jackson, MD, JD, Principal Investigator — Rutgers/NJMS
Locations (1):
- University Hospital, Newark, New Jersey, United States